CLINICAL TRIAL: NCT02948751
Title: Pilot Study Evaluating the Utility of OncoCEE (Cell Enrichment and Extraction) Technology, a Novel Immunocytochemical Microfluidic Device, in the Diagnosis of Leptomeningeal Metastasis (LM) From Breast Cancer Through Identification of Circulating Tumor Cells (CTCs) in Cerebrospinal Fluid (CSF)
Brief Title: Microfluidic Device to Diagnose Leptomeningeal Metastasis in Breast Cancer
Status: Completed | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Biocept, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAQ4761; R03CA208547-01 (NIH)
Record Dates: First submitted 2016-10-27; First posted 2016-10-28 (Estimated); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Leptomeningeal Metastasis
Keywords: Breast Carcinoma; Breast tumors; Cancer of the Breast; Malignant tumor of the breast; breast cancer; leptomeningeal metastasis
MeSH Terms: conditions — Breast Neoplasms; Meningeal Carcinomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (1):
- OncoCEE (Experimental): Patients with breast cancer who are undergoing lumbar puncture for suspicion of leptomeningeal metastasis. An additional CSF sample will be obtained for evaluation of CSF CTCs by OncoCEETM technology and cell-free DNA (recommended amount: 1 tube, 10 mL) at the time of lumbar puncture.
  Interventions: Device: OncoCEE

INTERVENTIONS:
Device: OncoCEE — The CSF sample will be to delivered to Biocept's laboratory for processing, and it will be evaluated for CTCs using OncoCEETM microchannel technology. This CSF sample will also be tested for cell-free circulating tumor DNA (ctDNA).
  Other Names: OncoCEETM microchannel technology

SUMMARY:
This study will prospectively enroll 36 evaluable subjects with breast cancer who are undergoing workup for clinical suspicion of leptomeningeal metastasis (LM). Neuroimaging consisting of MRI of the brain or total spine (or both, as clinically indicated) will be obtained in all patients. Patients will also undergo a lumbar puncture and standard CSF evaluation, which may consist of intracranial pressure measurement, CSF protein, glucose, white and red cell analysis, infectious cultures, as well as conventional cytopathologic analysis (cytocentrifuge). An additional CSF sample will be obtained for evaluation of CSF CTCs by OncoCEETM technology and cell-free DNA (recommended amount: 1 tube, 10 mL) at the time of lumbar puncture.

DETAILED DESCRIPTION:
Leptomeningeal metastasis (LM) is a condition in which cancer cells seed the meninges and may go on to invade the brain parenchyma, spinal cord, cranial nerves or peripheral nerves. It is a devastating complication of breast cancer, and is often considered in the differential diagnosis when patients with breast cancer present with new neurologic symptoms. It was previously thought to be a rare occurrence, but autopsy series have shown the true overall incidence to be up to 8%. In fact, while the incidence of meningeal metastasis from other malignancies has decreased, the opposite is true of breast cancer, in which clinical evidence suggests an increasing incidence.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older) patients, with invasive breast cancer, of all racial and ethnic origins
* Undergoing lumbar puncture for clinical or radiographic suspicion of leptomeningeal metastasis
* Provide study-specific informed consent
* Patients with unequivocal or suspicious MRI findings.
* Of those with a definitive diagnosis of LM (i.e. positive CSF cytology), 10 evaluable patients will be accrued.

Exclusion Criteria:

* Prior CSF fluid which identified malignant cells after 10 evaluable patients with positive CSF are accrued.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
In order to fulfill the requirement of sharing the data obtained in the research program, a website where the data acquired will be made available to the scientific community. Through this website, colleagues from other research centers will be able to read about the general information of the proposal, including its objectives and aims. The website will be updated on a regular basis (at least quarterly) to include the advances achieved during the research activities and new results obtained from data processing and statistical analysis. Hyperlinks pointing to other web pages with information related to the program will also be available on our website. These hyperlinks will be divided in those with information for patients and those with information for researchers.
  "briefly describe what specific individual participant data sets are to be shared (for example, all collected IPD, all IPD that underlie results in a publication)."
Time Frame: "A description of when the IPD and any additional supporting information will become available and for how long, including the start and end dates or period of availability. This may be provided as an absolute date (for example, starting in January 2025) or as a date relative to the time when summary data are published or otherwise made available (for example, starting 6 months after publication)."
Access Criteria: "Describe by what access criteria IPD and any additional supporting information will be shared, including with whom, for what types of analyses, and by what mechanism. Information about who will review requests and criteria for reviewing requests may also be provided."

REFERENCES:
- See also: Herbert Irving Comprehensive Cancer Center (HICCC) Clinical Trials Page — http://hiccc.columbia.edu/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OncoCEE
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OncoCEE
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Participants With Leptomeningeal Metastasis Detected (ER Status)
Description: Total number of participants with leptomeningeal metastasis detected (ER status)
Time Frame: 6 months
Population: Only includes patients with metastatic breast cancer enrolled with matched samples.
Measure: Count of Participants; unit: Participants
Arm/Group | OncoCEE
Number analyzed (Participants) | 11
Participants
  Detected by OncoCEE | 3
  Detected by standard lumbar puncture | 1

2. Primary Outcome: Total Number of Participants With Leptomeningeal Metastasis Detected (HER2 Status)
Description: Total number of participants with leptomeningeal metastasis detected (HER2 status)
Time Frame: 6 months
Population: Only includes patients with metastatic breast cancer enrolled with matched samples.
Measure: Count of Participants; unit: Participants
Arm/Group | OncoCEE
Number analyzed (Participants) | 11
Participants
  Detected by OncoCEE | 0
  Detected by standard lumbar puncture | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | OncoCEE
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT02948751/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT02948751/ICF_002.pdf